CLINICAL TRIAL: NCT02261402
Title: Effectiveness of "Medisinstart" - an Open Randomized Controlled Trial of a Newly Developed Pharmacy Service
Brief Title: Effectiveness of "Medisinstart"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apokus AS (Other)
Collaborators: Norwegian Pharmacy Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Apokus-001
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Cardiovascular Diseases
Keywords: Adherence; Morisky Medication Adherence Scale; Beliefs about Medicines Questionnaire; Medication Possession Ratio; Medication-Related Problems; Pharmacist; Pharmacist Intervention; Pharmacy; Pharmacy Service; Pharmacy Practice; Hypertension; Antihypertensive Agents; Anticoagulants; Statins; Dyslipidemia
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medisinstart (Experimental): Patients in this arm will receive the service; Medisinstart
  Interventions: Other: Medisinstart
- Current Practice (No Intervention): Patients in this arm will receive the current pharmacy practice of advice and guidance with their new medicine. This involves dispensing the medicine and briefly providing information regarding its use and potential side-effects.

INTERVENTIONS:
Other: Medisinstart — "Medisinstart" is a newly developed pharmacy service for patients about to start a new medicine for a chronic or long-term condition. It consists of two follow-up consultations with a pharmacist. The first at 1-2 weeks and the second at 3-5 weeks after start of the new medicine.
  Arms: Medisinstart

SUMMARY:
"Medisinstart" is a new service developed for use in Norwegian pharmacies. It is intended for patients that are about to start a new medicine for a chronic or long-term condition. It is based on research showing that problems with newly prescribed medicines appear rapidly and that a significant portion of patients quickly becomes non-adherent. The service consists of two follow-up consultations with a pharmacist. The first at 1-2 weeks and the second at 3-5 weeks after start of the new medicine.

The main purpose of this study is to investigate whether "Medisinstart" increases patients' adherence to the prescribed medication. Patients' beliefs about their medicines and their motivation for adherence will also be examined. The study also aims at revealing if "Medisinstart" has additional benefits for the patient, the society and the pharmacies.

ELIGIBILITY:
Inclusion Criteria:

First time prescription for a drug belonging to one of the following groups (ATC-code):

* Dabigatran etexilate (B01AE07)
* Rivaroxaban (B01AF01)
* Apixaban (B01AF02)
* Beta blocking agents (C07)
* Calcium channel blockers (C08)
* Agents acting on the renin-angiotensin system (C09)
* HMG CoA reductase inhibitors (statins) (C10AA)

Exclusion Criteria:

* Prior use (within the last 3 years) of the drug in question independent of strength, dose and formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1480 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Adherence by Morisky 8-item Medication Adherence Scale (MMAS-8) at 7 weeks | 7 weeks after dispensing the new medicine
  Adherence will be measured by a validated Norwegian translation of the MMAS-8
Adherence by Morisky 8-item Medication Adherence Scale (MMAS-8) at 18 weeks | 18 weeks after dispensing the new medicine
  Adherence will be measured by a validated Norwegian translation of the MMAS-8

SECONDARY OUTCOMES:
Self reported adherence at 7 weeks | 7 weeks after dispensing the new medicine
  Adherence will be measured by a Norwegian translation of the question: "People often miss taking doses of their medicines, for a wide range of reasons. Have you missed any doses of your new medicine the last week?"
Adherence by Medication Possession Ratio (MPR) at 18 weeks | 18 weeks after dispensing the new medicine
  Adherence by MPR will be calculated from data collected from the Norwegian Prescription Database
Patients' beliefs about their medicines by Beliefs about Medicines Questionnaire (BMQ) at inclusion | At inclusion
  Patients' beliefs about their medicines will be measured by a validated Norwegian translation of the BMQ
Self reported adherence at 18 weeks | 18 weeks after dispensing the new medicine
  Adherence will be measured by a Norwegian translation of the question: "People often miss taking doses of their medicines, for a wide range of reasons. Have you missed any doses of your new medicine the last week?"
Adherence by Medication Possession Ratio (MPR) at 1 year | 1 year after dispensing the new medicine
  Adherence by MPR will be calculated from data collected from the Norwegian Prescription Database
Patients' beliefs about their medicines by Beliefs about Medicines Questionnaire (BMQ) at 7 weeks | 7 weeks after dispensing the new medicine
  Patients' beliefs about their medicines will be measured by a validated Norwegian translation of the BMQ
Patients' beliefs about their medicines by Beliefs about Medicines Questionnaire (BMQ) at 18 weeks | 18 weeks after dispensing the new medicine
  Patients' beliefs about their medicines will be measured by a validated Norwegian translation of the BMQ

OTHER OUTCOMES:
Number of reported Medication-Related Problems in the intervention arm | During the intervention
  The pharmacist carrying out the intervention will report all discovered Medication-Related Problems
Patients' evaluation of "Medisinstart" | 7 weeks after dispensing the new medicine
  Patients' in the intervention arm will evaluate the service by answering a questionnaire
Pharmacists' evaluation of patient benefit | 7 months after start of the study
  Pharmacists performing the service will answer the following question (translated from Norwegian): "You have currently performed "Medisinstart" with at least 5 patients. Do you regard it to be beneficial for the patients?"
Pharmacy costs by performing the service | 1 year after study start
  Pharmacies will report the COSTs for carrying out the service

CONTACTS AND LOCATIONS:
Overall Officials: Karine W Ruud, PhD, Study Director — Apokus AS; Sara Bremer, PhD, Study Director — Apokus AS; Ragnar Hovland, PhD, Study Director — Photocure ASA (current affiliation), Apokus AS (until Dec. 2016)
Locations (67):
- Norway (67):
  - Apotek 1 Alta, Alta
  - Apotek 1 Andselv, Andselv
  - Boots apotek Harebakken, Arendal
  - Sykehusapoteket Arendal, Arendal
  - Boots apotek Moa, Ålesund
  - Vitusapotek Raumnes, Årnes
  - Vitusapotek Årnes, Årnes
  - Apotek 1 Horisont, Bergen
  - Boots apotek Bryggen, Bergen
  - Sjukehusapoteket i Bergen, Bergen
  - Sykehusapoteket i Bodø, Bodø
  - Apotek 1 Brandbu, Brandbu
  - Apotek 1 Bømlo, Bremnes
  - Apotek 1 Åssiden, Drammen
  - Sykehusapoteket Drammen, Drammen
  - Boots apotek Elverum, Elverum
  - Sykehusapoteket Elverum, Elverum
  - Boots apotek Flisa, Flisa
  - Apotek 1 Helsehuset Fredrikstad, Fredrikstad
  - Sjukehusapoteket i Førde, Førde
  - Boots apotek Hamar, Hamar
  - Sjukehusapoteket i Haugesund, Haugesund
  - Apotek 1 Lerka, Kleppe
  - Apotek 1 Kopervik, Kopervik
  - Vitusapotek Sørlandssenteret, Kristiansand
  - Boots apotek Larvik, Larvik
  - Apotek 1 Lofotsenteret, Leknes
  - Apotek 1 Malvik, Malvik
  - Apotek 1 Mandal, Mandal
  - Ditt apotek Maura, Maura
  - Ditt apotek Meyer, Mo i Rana
  - Ditt apotek Ytteren, Mo i Rana
  - Apotek 1 Sjøsiden, Mosjøen
  - Vitusapotek Varnaveien Moss, Moss
  - Apotek 1 Morenen, Mysen
  - Vitusapotek Nesbru, Nesbru
  - Apotek 1 St. Hanshaugen senter, Oslo
  - Boots apotek Bogstadveien, Oslo
  - Boots apotek Skøyen, Oslo
  - Boots apotek Solli, Oslo
  - Diakonhjemmets sykehusapotek, Oslo
  - Lovisenberg sykehusapotek, Oslo
  - Sykehusapoteket Oslo, Ullevål, Oslo
  - Vitusapotek Storo, Oslo
  - Vitusapotek Raufoss, Raufoss
  - Apotek 1 Kvadrat, Sandnes
  - Vitusapotek Ganddal, Sandnes
  - Vitusapotek Syv Søstre, Sandnessjøen
  - Apotek 1 Sandvika Storsenter, Sandvika
  - Sykehusapoteket Bærum, Sandvika
  - Boots apotek Lande, Sarpsborg
  - Boots apotek Saupstad, Saupstad
  - Vitusapotek Selbak, Sellebakk
  - Apotek 1 Ski Amfi, Ski
  - Sykehusapoteket Skien, Skien
  - Apotek 1 Hjorten Stavanger, Stavanger
  - Sjukehusapoteket i Stavanger, Stavanger
  - Vitusapotek Løven Stavanger, Stavanger
  - Vitusapotek Medisinsk senter - Steinkjer, Steinkjer
  - Sykehusapoteket Lørenskog, Strømmen
  - Vitusapotek Strømmen storsenter, Strømmen
  - Vitusapotek K1 Tromsø, Tromsø
  - Boots apotek Nordre, Trondheim
  - Vitusapotek Solsiden, Trondheim
  - Sykehusapoteket Tønsberg, Tønsberg
  - Vitusapotek Innherred, Verdal
  - Gausdal apotek, Østre Gausdal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barber N, Parsons J, Clifford S, Darracott R, Horne R. Patients' problems with new medication for chronic conditions. Qual Saf Health Care. 2004 Jun;13(3):172-5. doi: 10.1136/qhc.13.3.172. PMID 15175485
- [Background] Boyd M, Waring J, Barber N, Mehta R, Chuter A, Avery AJ, Salema NE, Davies J, Latif A, Tanajewski L, Elliott RA. Protocol for the New Medicine Service Study: a randomized controlled trial and economic evaluation with qualitative appraisal comparing the effectiveness and cost effectiveness of the New Medicine Service in community pharmacies in England. Trials. 2013 Dec 1;14:411. doi: 10.1186/1745-6215-14-411. PMID 24289059
- [Background] Clifford S, Barber N, Elliott R, Hartley E, Horne R. Patient-centred advice is effective in improving adherence to medicines. Pharm World Sci. 2006 Jun;28(3):165-70. doi: 10.1007/s11096-006-9026-6. Epub 2006 Sep 27. PMID 17004019
- [Background] Elliott RA, Barber N, Clifford S, Horne R, Hartley E. The cost effectiveness of a telephone-based pharmacy advisory service to improve adherence to newly prescribed medicines. Pharm World Sci. 2008 Jan;30(1):17-23. doi: 10.1007/s11096-007-9134-y. Epub 2007 Jun 8. PMID 17557211
- [Background] Haynes RB, McDonald H, Garg AX, Montague P. Interventions for helping patients to follow prescriptions for medications. Cochrane Database Syst Rev. 2002;(2):CD000011. doi: 10.1002/14651858.CD000011. PMID 12076376
- [Background] Horne R, Weinman J. Patients' beliefs about prescribed medicines and their role in adherence to treatment in chronic physical illness. J Psychosom Res. 1999 Dec;47(6):555-67. doi: 10.1016/s0022-3999(99)00057-4. PMID 10661603
- [Background] Hov I, Bjartnes M, Slordal L, Spigset O. [Are drugs taken as prescribed?]. Tidsskr Nor Laegeforen. 2012 Feb 21;132(4):418-22. doi: 10.4045/tidsskr.11.0225. Norwegian. PMID 22353834
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Ruths S, Viktil KK, Blix HS. [Classification of drug-related problems]. Tidsskr Nor Laegeforen. 2007 Nov 29;127(23):3073-6. Norwegian. PMID 18049498
- [Background] Sabate E. (Ed.) (2003), Adherence to Long-Term Therapies: Evidence for Action. Geneva, Switzerland: World Health Organization